CLINICAL TRIAL: NCT06478433
Title: "Efficacy and Safety Study of the Medical Device Munatoril® Aerosol Combo in the Recovery of Nasal Homeostasis in Pediatric Patients Undergoing Adenoidectomy or Adenotonsillectomy."
Brief Title: Study on the Efficacy and Safety of a Device for Post-op Recovery in Pediatric Adenectomy/Adenotonsillectomy.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmaluce srl (Industry)
Collaborators: Gruppo FarmaImpresa (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Munatoril® Aerosol Combo_2024
Record Dates: First submitted 2024-06-26; First posted 2024-06-27 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Adenoidal Disorder; Tonsillitis; Otorhinolaryngologic Diseases; Nasal Disease
Keywords: nasal irrigation
MeSH Terms: conditions — Tonsillitis; Otorhinolaryngologic Diseases; Nose Diseases

STUDY DESIGN:
Intervention Model Description: Prospective prospective single-center controlled non-randomized for-profit interventional study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Munatoril (Experimental): Experimental: Munatoril From day 1 to day 7 postoperatively: SID administration of Munatoril® Aerosol Combo by aerosol therapy, in the morning + TID administration of an over-the-counter sterile isotonic solution by Lavonase® syringe.
  From day 8 to day 14 postoperatively:
  SID administration of Munatoril® Aerosol Combo via Lavonase® syringe, in the morning + TID administration of an over-the-counter sterile isotonic solution, via Lavonase® syringe.
  - From postoperative day 15 to day 29: TID administration via Lavonase® syringe of an isotonic solution obtained by diluting Munatoril® Aerosol Combo hypertonic solution
  Interventions: Device: Munatoril Aerosol Combo
- Control (Active Comparator): Active Comparator: Control Day 1 to day 7 postoperative: SID administration of Hypertonic Solution by aerosol therapy, in the morning + TID administration of an over-the-counter sterile isotonic solution by Lavonase® syringe.
  Postoperative day 8 to day 14:
  SID administration of hypertonic solution via Lavonase® syringe, in the morning + TID administration of an over-the-counter sterile isotonic solution, via Lavonase® syringe.
  - Postoperative day 15 to day 29: TID administration via Lavonase® syringe of an isotonic solution.
  Interventions: Device: Iperclenny

INTERVENTIONS:
Device: Munatoril Aerosol Combo — Munatoril® Aerosol Combo is a Medical Device that contains:
  5 ml single-dose vials of sterile, 3% hypertonic, near-neutral pH bromine-iodine saline solution, based on Cervia integral sea salt, salso-bromo-iodine saline mother water from the Cervia Thermal Baths and hyaluronic acid with high molecular weight.
  Lavonase® syringe with blue nebulizer valve (microsol), 10 ml, Medical Device for the administration of solutions in nebulized form within the nasal cavities and nasopharynx.
  Arms: Munatoril
Device: Iperclenny — Hypertonic and Isotonic solution present on market in italy.
  Other Names: Isoclenny
  Arms: Control

SUMMARY:
The objective of this prospective pre-market interventional clinical study is to evaluate the efficacy and safety of the medical device Munatoril® Aerosol Combo in its different modalities of use, through the analysis of clinical and subjective outcomes in children operated on adenoidectomy or adenotonsillectomy, compared with a hypertonic solution and an over-the-counter isotonic solution (control group).

The primary question it aims to answer is whether the components prensent in Munatoril provide a benefit and whether they play a role in the recovery of nasal homeostasis following adeinodectomy and adenotonsillectomy compared with an over-the-counter hypertonic saline solution.

Endpoints Evaluation of subjective longitudinal differences (intragroup over-time change) and differences between study group and control group (intergroup difference) regarding the use of the medical device, obtained following the protocol, with assessment at 8, 15 and 30 days after surgery by Likert Scale Score for tolerability, and at 0, 15 and 30 days by SNOT22 Score and Lund-Kennedy Endoscopic Score for efficacy.

In addition, there is a recording of any adverse events in both groups at 8, 15 and 30 days post-surgery, and an inter-group comparative evaluation.

Participants: Pediatric patients who are candidates for adenoidectomy or adenotonsillectomy surgery at the study site facility will be systematically evaluated preoperatively for inclusion in the clinical trial and possibly recruited. Follow-up will last 30 days.

DETAILED DESCRIPTION:
Sample selection criteria

Inclusion criteria.

Patients of either sex aged 2 to 17 years, candidates for adenoidectomy or adenotonsillectomy surgery.

Acquisition and signing of informed consent by the legal guardian. Exclusion criteria.

Syndromic patients. Patients allergic to any substance in the study formulations. Patients who have used intranasal corticosteroids, topical or systemic corticosteroids, or any intranasal medication in the week prior to study entry.

Active respiratory infection in the 2 weeks prior to study entry. Patients with a history of chronic epistaxis or immunodeficiency. 2.3 Study exit criteria.

For reasons related to study treatment (adverse event); for reasons related to surgery (adverse event); for non-treatment-related reasons (death due to illness, patient transfer to other treatment site); for patient-related reasons (withdrawal of consent, poor compliance); for reasons related to compliance with procedures/other (protocol violations, administrative problems); for withdrawal of consent by the patient's parents or legal guardians. In cases of exit from follow-up, there is provision for reporting the exit, including the date and reasons for it.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex aged 2 to 17 years who are candidates for adenoidectomy or adenotonsillectomy surgery.
* Acquisition and signing of informed consent by the legal guardian.

Exclusion Criteria:

* Syndromic patients.
* Patients allergic to any substance in the study formulations.
* Patients who have used intranasal corticosteroids, topical or systemic corticosteroids, or any intranasal medication in the week prior to study entry.
* Active respiratory infection in the 2 weeks prior to study entry.
* Patients with a history of chronic epistaxis or immunodeficiency.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Subjective evaluation for efficacy: QoL | T0 (preoperative) - T2 (15 days) - T3 (30 days).
  The investigator will use the questionnaire "Sino-Nasal Outcome Test-22 (SNOT-22)" for the evaluation of QoL and the symptoms impact on patient's life. The SNOT-22 is based on a Likert scale where 0 = "No problem", 1 = "Very mild problem", 2 = "Mild or slight problem", 3 = "Moderate problem", 4 = "Severe problem", and 5 = "Problem as bad as it can be." Are 22 items and the score can be from 0 to 110. Higher scores means a worse outcome.

SECONDARY OUTCOMES:
Objective evaluation for efficacy: Lund-kennedy Score | T0 (intraopertory ) - T2 (15 days) - T3 (30 days).
  Lund-kennedy Score: This score assesses the severity of three objective data trough nasal endoscopy. It is polyps (0, none; 1, in the middle meatus; 2, beyond the middle meatus); discharge (0, none; 1, clear and thin; 2, thick and purulent); edema (0, absent; 1, mild; 2, severe); scarring/adhesions (0, absent; 1, mild; 2, severe); and crusting (0, absent; 1, mild; 2, severe). The score can be from 0 to 10. Higher scores means a worse outcome.

OTHER OUTCOMES:
Tolerability and recording of any adverse events to assess safety profile | T1 (8 days - telephone administration) - T2 (15 days) - T3 (30 days).
  Likert Scale Score from 1 to 5 score. Higher scores means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Tedeschi, Master, Study Chair — Gruppo FarmaImpresa

IPD SHARING:
Plan to Share IPD: No